CLINICAL TRIAL: NCT02968459
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cell Local Intramuscular Injection for Treatment of Uterine Scars
Brief Title: Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cell Local Intramuscular Injection for Treatment of Uterine Scars
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The pandemic resulted in no enrollments.
Sponsor: Maternal and Child Health Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Zhengping Liu, MD, Director, Maternal and Child Health Hospital of Foshan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCHHFoshan-1603
Record Dates: First submitted 2016-11-14; First posted 2016-11-18 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Uterine Scar
Keywords: Mesenchymal Stem Cells; Cesarean Section; Uterine Scar
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical cord MSCs Group (Experimental): 1*10^7 Umbilical cord MSCs
  Interventions: Other: Umbilical cord MSCs
- Placebo-Controlled Group (Placebo Comparator): 1ml of 0.9% saline
  Interventions: Other: 0.9% Saline

INTERVENTIONS:
Other: Umbilical cord MSCs — Participants will receive direct local intramuscular injection of 1*10^7 MSCs (in 1ml of 0.9% saline) in the uterine incision.
  Arms: Umbilical cord MSCs Group
Other: 0.9% Saline — Participants will receive direct local intramuscular injection 1ml of 0.9% saline in the uterine incision.
  Arms: Placebo-Controlled Group

SUMMARY:
This is a single center, randomized, double blind, placebo controlled study to evaluate the safety and efficacy of umbilical cord mesenchymal stem cell local intramuscular injection for treatment of caesarean section uterine scars.

DETAILED DESCRIPTION:
In recent decades, the percentage of Cesarean section (CS) deliveries has dramatically increased around the world. While it allows safe delivery in many situations, the risks of severe maternal complications associated with cesarean delivery are higher than those associated with vaginal delivery. These maternal complications include short term, long-term, the next pregnancy, and the non-pregnant state, such as abnormal uterine bleeding and postmenstrual spotting.

Uterine niche, also named cesarean scar defect, deficient cesarean scar, pouch, or diverticulum, is defined as a triangular anechoic structure at the site of the scar or a gap in the myometrium at the site of a previous caesarean section. It is one of the most common complications associated with previous cesarean section. The primary clinical manifestation is postmenstrual spotting, which may seriously affect the daily life of patients. The treatment includes medical treatment, such as oral contraceptives, and surgical methods, such as hysteroscopy resectoscopic correction, endometrial ablation, laparoscopic surgery, and transvaginal repair surgery. Although good outcomes are reported in each study, present treatments could not decrease the incidence among women after undergoing cesarean section.

Mesenchymal stem cells (MSCs) are long-lived cells with the ability of both self-renewal and differentiation into multi-potential cells, such as osteoblasts, adipocytes and smooth muscle cells. Trials with MSCs in patients after myocardial infarction have shown an excellent safety and efficacy. In this trial, the investigators postulate that MSCs can reduce uterine niche and convert scar tissue to viable myometrium. To test the hypothesis, the investigators therefore undertake a Phase II clinical trial of the treatment for uterine niche among primiparous women who undergo cesarean section.

This is a randomized, double-blind, placebo-controlled clinical trial designed to investigate the efficacy and safety of umbilical cord mesenchymal stem cells treatment on the caesarean section uterine scars. A total of one hundred and twenty (120) participants will be randomized (1:1) to receive direct local intramuscular injection of 1*10^7 MSCs (a dose of 1*10^7 cells in 1 ml of 0.9% saline) (MSCs group) or an identical-appearing 1ml of 0.9% saline placebo (placebo-controlled group). Cesarean procedures and care will follow usual practices. All participants will be performed by obstetricians from the investigators' department using a unified double-layer uterine closure technique with a continuous absorbable polyglycolic 1-0 suture. After suturing the uterine incision, direct local intramuscular injection will be performed in the uterine incision as soon as possible on the operating table. One ml solution will be injected as twenty aliquots of 0.05ml into each injection site on the incision. Injection sites will be selected near the incision at evenly 20 different sites. Participants will be followed up at 6 weeks, 3 months and 6 months. For the purpose of the endpoint analysis and safety evaluations, the investigators will utilize an "intention-to-treat" study population.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women receiving cesarean delivery
* Ages between 21-35 years
* Gestation ages ≥ 37 weeks and < 42 weeks
* Willing to comply with study dosing and completed the entire course of the study
* Willing to give and sign an informed consent form and a photographic release form

Exclusion Criteria:

* Fibroids
* Placenta previa
* Placenta abruption
* Multiple gestation
* Antepartum hemorrhage
* Preeclampsia/Eclampsia
* Hepatic or renal dysfunction
* Any systemic uncontrolled disease
* Inability to provide consent

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with uterine niche | 6 months post treatment
  The niche is defined as a triangular anechoic area at the presumed site of incision in the uterus by transvaginal utrasonography.

SECONDARY OUTCOMES:
Change of uterine scar thickness | 6 weeks, 3 and 6 months post treatment
  The scar thickness be measured using a transvaginal utrasonography
Change of uterine scar area | 6 weeks, 3 and 6 months post treatment
  The scar area will be measured using a transvaginal utrasonography
Number of participants with endometritis | 6 months post treatment
  Endometritis is defined as the presence of at least two of the following signs with no other recognized cause: fever (temperature of at least 38℃), abdominal pain, uterine tenderness, or purulent drainage from the uterus.
Number of participants with wound infection | 6 months post treatment
  Wound infection is defined as the presence of either superficial or deep incisional surgical-site infection characterized by cellulitis or erythema and induration around the incision or purulent discharge from the incision site with or without fever and included necrotizing fasciitis.
Immunoglobulin concentrations in breast milk and serum | 6 weeks, 3 and 6 months post treatment
  Breast milk and serum immunoglobulin (IgG, IgA, IgM) and the complement (C3, C4) are detected by transmission immune turbidity method using automatic biochemical analyzer.
Adverse events occurrence | 6 months post treatment
  Adverse events will be evaluated since the baseline visit until 6 months after the end of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengping Liu, MD, Principal Investigator — Maternal and Child Health Hospital of Foshan
Locations (1):
- Maternal and Child Health Hospital of Foshan, Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fan D, Wu S, Ye S, Wang W, Guo X, Liu Z. Umbilical cord mesenchyme stem cell local intramuscular injection for treatment of uterine niche: Protocol for a prospective, randomized, double-blinded, placebo-controlled clinical trial. Medicine (Baltimore). 2017 Nov;96(44):e8480. doi: 10.1097/MD.0000000000008480. PMID 29095305